CLINICAL TRIAL: NCT03511937
Title: A Randomized Controlled Trial Evaluating the Impact of Sugar-Sweetened Beverage Health Warnings on Purchases
Brief Title: Impact of Sugar-Sweetened Beverage Health Warnings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: North Carolina Translational and Clinical Sciences Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 17-3375; 2KR951708 (Other Grant/Funding Number: North Carolina Translational and Clinical Sciences Institute)
Record Dates: First submitted 2018-04-18; First posted 2018-04-30 (Actual); Results first posted 2021-03-10 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: Dietary Habits
Keywords: Food and beverage purchases; Sugar-sweetened beverages; Beverages
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Who Masked: Participant
Masking Description: This trial uses incomplete disclosure to mask the purpose of the trial from participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sugar-Sweetened Beverage Health Warning Label (Experimental)
  Interventions: Behavioral: Sugar-Sweetened Beverage Health Warning Label
- Neutral Label (Other)
  Interventions: Other: Neutral Label

INTERVENTIONS:
Behavioral: Sugar-Sweetened Beverage Health Warning Label — Labels with a health warning will be applied to the front-of-package of all sugar-sweetened beverage containers in the mock store. Investigators developed the text and design of these labels based on previous research and on designs described in US and international legislation.
  Arms: Sugar-Sweetened Beverage Health Warning Label
Other: Neutral Label — Neutral labels will be applied to the front-of-package of all sugar-sweetened beverage containers in the mock store. Investigators developed the design of these labels.
  Arms: Neutral Label

SUMMARY:
Consumption of sugar-sweetened beverages (SSBs) like sodas, sports drinks, and fruit drinks remains a pressing public health concern in the United States. Consumption of SSBs remains well above recommended levels, and has been linked to obesity, diabetes, and cardiovascular disease. In response, policymakers across the U.S. have proposed requiring warning messages on SSB containers to inform the public and reduce consumption to healthier levels. While online studies find that such warnings reduce intentions to purchase SSBs, no studies have yet examined the impact of warnings on actual consumer behavior. The purpose of this randomized trial is to determine whether health warnings on sugar-sweetened beverages are more effective than control labels at reducing purchases of sugar-sweetened beverages. The trial will take place in a mock convenience store. Participants will be randomly assigned to a health warnings arm in which all sugar-sweetened beverages in the store are labeled with a health warning, or to a control arm in which all sugar-sweetened beverages in the store are labeled with a neutral label. Participants will select items to purchase with cash, and purchases will be compared across trial arms.

DETAILED DESCRIPTION:
Background: Obesity, diabetes and cardiovascular disease are among the leading causes of death in the United States. Consumption of sugar-sweetened beverages (SSBs) such as sodas, fruit drinks and sports drinks increases risk of these preventable conditions. SSBs are particularly problematic because they are high in calories but offer little nutritional value, and because the liquid calories in SSBs cause faster spikes in blood sugar and lower feelings of fullness than solid foods.

Despite these risks, the average American adult consumes more than 130 calories per day from SSBs, well above recommended levels. A promising strategy for reducing SSB consumption is requiring health warnings on SSB containers. Online studies show that health warnings attract consumers' attention and reduce intentions to purchase SSBs. However, no research has tested the impact of SSB health warnings on actual behaviors. This randomized trial evaluates whether health warnings reduce purchases of SSBs.

Setting: The trial will take place a mock convenience store setting created for researchers to examine how store and product characteristics influence consumer purchases in a controlled but realistic environment. The store reflects a convenience store's characteristics, selling foods, beverages, and household items at real-world prices. Participants can buy these products using cash.

Recruitment: Participants will be recruited via university community subject pools, printed flyers posted, and online listings. Interested potential participants will complete an online pre-enrollment screening questionnaire to determine their eligibility. If eligible, they will be invited to schedule a time to visit the mock store for the trial.

Informed consent: At the beginning of the study visit, research staff will review the consent documents with the participants. After reviewing the form, the research staff member will ask the participant if he or she has any questions. Then both parties will sign the consent form and the participant will receive a copy of the consent form to keep.

Randomization: Participants will be randomly assigned to trial arms. An independent biostatistician will conduct the randomization a priori. Participants will have an equal chance of being randomized to either arm of the trial. Randomization will be carried out by generating a random number for each participant identification code (ID). Participant IDs will be ordered on this random number from smallest to largest. The bottom half of the IDs will be assigned to the control arm and the top half to the treatment arm (trial arms are described below). When participants arrive for their study visit, they will be assigned the next consecutive participant ID and will be allocated to the trial arm previously assigned to that ID.

Experimental Procedures: When participants arrive at the mock store, they will be provided with a shopping basket and their participation incentive in cash. Participants will be instructed to pretend they are on a usual shopping trip and reminded that there are no right or wrong products to select. They will not be told the trial's purpose.

Participants will be asked to complete a shopping task. They will be given a list of product categories and asked to select their preferred products in each of these categories. They will indicate their selections by placing products in their shopping basket. Before they begin the shopping task, participants will be instructed that they will be required to purchase one of the items they select, and that this item will be chosen for them at random by the experimenter. This procedure incentivizes participants to only select products they are actually interested in purchasing. After participants have completed the shopping task, the experimenter will randomly choose one of the products in the participant's basket for participant to purchase with his or her incentive cash. The participant will pay for the product and will receive change as necessary. After paying for their item, participants will complete a computer-based survey in another room.

Assessment: The products participants select will be recorded by the experimenter at the end of the shopping task. Participants will also complete 1 computer-based survey immediately after completing the shopping task.

Detailed description of the trial arms: Participants will be assigned to either a health warnings arm or a control arm. In the health warnings arm, all SSB products will be labeled with a health warning label. Investigators developed the text and design of these labels based on previous research and on label designs described in US and international legislation. In the control arm, all SSB products will be labeled with a neutral label, also developed by the investigators. In both arms, labels will be adhered directly on the front-of-package of SSB containers.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Consume at least 12oz/week of sugar-sweetened beverages during the past month
* Be able to read and speak English

Exclusion Criteria:

* Under the age of 18 years
* Consume less than 12 ounces/week of sugar-sweetened beverages during the past month
* Unable to read or speak English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2018-05-11 (Actual); Primary Completion 2018-09-19 (Actual); Study Completion 2018-09-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anna H Grummon, MSPH, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bollard T, Maubach N, Walker N, Ni Mhurchu C. Effects of plain packaging, warning labels, and taxes on young people's predicted sugar-sweetened beverage preferences: an experimental study. Int J Behav Nutr Phys Act. 2016 Sep 1;13(1):95. doi: 10.1186/s12966-016-0421-7. PMID 27580589
- [Background] Roberto CA, Wong D, Musicus A, Hammond D. The Influence of Sugar-Sweetened Beverage Health Warning Labels on Parents' Choices. Pediatrics. 2016 Feb;137(2):e20153185. doi: 10.1542/peds.2015-3185. Epub 2016 Jan 14. PMID 26768346
- [Background] Zoellner J, Estabrooks PA, Davy BM, Chen YC, You W. Exploring the theory of planned behavior to explain sugar-sweetened beverage consumption. J Nutr Educ Behav. 2012 Mar-Apr;44(2):172-7. doi: 10.1016/j.jneb.2011.06.010. Epub 2011 Dec 8. PMID 22154130
- [Background] Nonnemaker, J., Farrelly, M., Kamyab, K., Busey, A., & Mann, N. (2010). Experimental study of graphic cigarette warning labels. Final Results Report. RTI Project, 7. Accessed March 20, 2018. Available at: http://www.tobaccolabels.ca/wp/wp-content/uploads/2013/12/USA-2010-Experimental-Study-of-Graphic-Cigarette-Warning-Labels-Final-Results-Report-and-Appendices-FDA.pdf
- [Background] Moodie C, MacKintosh AM, Hammond D. Adolescents' response to text-only tobacco health warnings: results from the 2008 UK Youth Tobacco Policy Survey. Eur J Public Health. 2010 Aug;20(4):463-9. doi: 10.1093/eurpub/ckp199. Epub 2009 Dec 3. PMID 19959613
- [Background] Klein WM, Zajac LE, Monin MM. Worry as a moderator of the association between risk perceptions and quitting intentions in young adult and adult smokers. Ann Behav Med. 2009 Dec;38(3):256-61. doi: 10.1007/s12160-009-9143-2. PMID 20049660
- [Background] Fathelrahman AI, Omar M, Awang R, Cummings KM, Borland R, Bin Mohd Samin AS. Impact of the new Malaysian cigarette pack warnings on smokers' awareness of health risks and interest in quitting smoking. Int J Environ Res Public Health. 2010 Nov;7(11):4089-99. doi: 10.3390/ijerph7114089. Epub 2010 Nov 22. PMID 21139879
- [Background] Brewer NT, Jeong M, Mendel JR, Hall MG, Zhang D, Parada H Jr, Boynton MH, Noar SM, Baig SA, Morgan JC, Ribisl KM. Cigarette pack messages about toxic chemicals: a randomised clinical trial. Tob Control. 2019 Jan;28(1):74-80. doi: 10.1136/tobaccocontrol-2017-054112. Epub 2018 Apr 13. PMID 29654122
- [Derived] Grummon AH, Taillie LS, Golden SD, Hall MG, Ranney LM, Brewer NT. Sugar-Sweetened Beverage Health Warnings and Purchases: A Randomized Controlled Trial. Am J Prev Med. 2019 Nov;57(5):601-610. doi: 10.1016/j.amepre.2019.06.019. Epub 2019 Oct 2. PMID 31586510

RESULTS

PARTICIPANT FLOW:
Groups:
- Sugar-Sweetened Beverage (SSB) Health Warning Label: Labels with a health warning will be applied to the front-of-package of all sugar-sweetened beverage (SSB) containers in the mock store. Investigators developed the text and design of these labels based on previous research and on designs described in US and international legislation.
Period: Overall Study
Arm/Group | Sugar-Sweetened Beverage (SSB) Health Warning Label | Neutral Label
Started | 200 | 200
Completed | 200 | 200
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sugar-Sweetened Beverage Health Warning Label | Neutral Label | Total
Number analyzed (Participants) | 200 | 200 | 400
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.0 (10.5) | 29.0 (10.3) | 29.0 (10.3)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 76 | 83 | 159
  Female | 121 | 115 | 236
  Transgender or other | 3 | 2 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 25 | 34
  Not Hispanic or Latino | 191 | 175 | 366
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 51 | 47 | 98
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
  Black or African American | 43 | 46 | 89
  White | 93 | 87 | 180
  More than one race | 5 | 12 | 17
  Unknown or Not Reported | 5 | 8 | 13
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 200 | 200 | 400

OUTCOME MEASURES:

1. Primary Outcome: Mean Number of Calories (kcal) Purchased From Sugar-sweetened Beverages
Description: The primary outcome is calories of sugar-sweetened beverages purchased during the shopping task. Calories from sugar-sweetened beverage purchases is defined as the total number of calories from sugar-sweetened beverages in the participant's basket when they complete the shopping task, calculated as the sum of calories/container for all SSB containers. Purchases will be recorded by the experimenter immediately after the participant completes the ~10-minute shopping task.
Time Frame: At completion of ~10-minute shopping task
Measure: Mean (Standard Deviation); unit: kcal
Arm/Group | Sugar-Sweetened Beverage Health Warning Label | Neutral Label
Number analyzed (Participants) | 200 | 200
kcal | 109.9 (134.9) | 143.2 (137.4)
Statistical Analysis 1: Comparison: Sugar-Sweetened Beverage Health Warning Label vs Neutral Label; Test type: Superiority; p = 0.02, Two-part regression model with robust SE — The a priori threshold for statistical significance was < 0.05; Analyses controlled for overweight/obese status and Hispanic ethnicity, which were unbalanced between arms, and estimated Huber-White robust SEs; Mean Difference (Final Values) = -31.4, 95% CI 2-sided [-57.9 to -5.0]

2. Secondary Outcome: Mean Number of Calories (kcal) Purchased From All Foods and Beverages
Description: Total calories purchased from all foods and beverages is defined as the total number of calories from all products (including sugar-sweetened beverages, non-sugar-sweetened beverages, and all foods) in the participant's basket when they complete the shopping task. Total calories purchased will be calculated as the sum of calories/container for all products. Purchases will be recorded by the experimenter immediately after the participant completes the ~10 minute shopping task.
Time Frame: At completion of ~10-minute shopping task
Measure: Mean (Standard Deviation); unit: kcal
Arm/Group | Sugar-Sweetened Beverage Health Warning Label | Neutral Label
Number analyzed (Participants) | 200 | 200
kcal | 2365.6 (1172.4) | 2435.6 (1095.7)
Statistical Analysis 1: Comparison: Sugar-Sweetened Beverage Health Warning Label vs Neutral Label; Test type: Superiority; p = 0.55, Regression, Linear — The a priori threshold for statistical significance was < 0.05; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -69.4, 95% CI 2-sided [-295.5 to 156.6]

3. Secondary Outcome: Percent of Participants Who Purchase a Sugar-sweetened Beverage
Description: Purchase of a sugar-sweetened beverage is defined as the participant having one or more sugar-sweetened beverage in their basket when they complete the shopping task. Purchases will be recorded by the experimenter immediately after the participant completes the ~10-minute shopping task.
Time Frame: At completion of ~10-minute shopping task
Measure: Number; unit: percentage of participants
Arm/Group | Sugar-Sweetened Beverage Health Warning Label | Neutral Label
Number analyzed (Participants) | 200 | 200
percentage of participants | 50.0 | 64.0
Statistical Analysis 1: Comparison: Sugar-Sweetened Beverage Health Warning Label vs Neutral Label; Test type: Superiority; p = 0.006, Regression, Logistic — The a priori threshold for statistical significance was < 0.05; Analyses controlled for overweight/obesity status and Hispanic ethnicity, which were unbalanced between treatment arms; Mean Difference (Final Values) = -13, 95% CI 2-sided [-23 to -4] — Analyses used logistic regression to calculate mean difference in predicted probability of purchasing a sugar-sweetened beverage

4. Secondary Outcome: Mean Number of Sugar-sweetened Beverages Purchased
Description: Number of sugar-sweetened beverages purchased is defined as the number of sugar-sweetened beverages in the participants' basket when they complete the shopping task. Purchases will be recorded by the experimenter immediately after the participant completes the ~10-minute shopping task.
Time Frame: At completion of ~10 minute shopping task
Measure: Mean (Standard Deviation); unit: Beverages
Arm/Group | Sugar-Sweetened Beverage Health Warning Label | Neutral Label
Number analyzed (Participants) | 200 | 200
Beverages | 0.7 (0.8) | 0.9 (0.8)
Statistical Analysis 1: Comparison: Sugar-Sweetened Beverage Health Warning Label vs Neutral Label; Test type: Superiority; p = 0.010, Negative binomial regression — The a priori threshold for statistical significance was < 0.05; Analyses controlled for overweight/obesity status and Hispanic ethnicity, which were unbalanced between arms, and estimated Huber-White robust SEs; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-0.4 to -0.1]

5. Secondary Outcome: Mean Intentions Score to Limit Consumption of Beverages Added Sugar
Description: Intentions to limit consumption of beverages with added sugar will be measured at post-test using 3 items adapted from Klein, Zajax & Monin (2009). The items ask participants to rate the extent to which they want to, plan to, and are likely to, drink less than 1 beverage with added sugar in the next week. Responses to these three items will be averaged to create a mean intentions score. Response options are on a 1 to 7 scale, thus, mean scores can range from 1-7, with higher scores indicating higher intentions to limit consumption of beverages with added sugar.
Time Frame: Within 30 minutes following completion of ~10-minute shopping task
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sugar-Sweetened Beverage Health Warning Label | Neutral Label
Number analyzed (Participants) | 200 | 200
score on a scale | 4.8 (1.8) | 4.7 (1.8)
Statistical Analysis 1: Comparison: Sugar-Sweetened Beverage Health Warning Label vs Neutral Label; Test type: Superiority; p = 0.403, Regression, Linear — The a priori threshold for statistical significance was < 0.05; Analyses controlled for obesity status and Hispanic ethnicity, which were unbalanced between arms, and estimated Huber-White robust standard errors; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [-0.2 to 0.5]

6. Secondary Outcome: Mean Intentions Sore to Limit Consumption of Specific Sugar-sweetened Beverages
Description: Intentions to limit consumption of specific beverage categories (i.e., soda, fruit drinks, sport drinks/flavored waters, sweetened coffee/tea, and energy drinks) will be measured at post-test using measures adapted from Klein, Zajax, & Monin (2009). For each of the five beverage categories, participants will rate the extent to which they are likely to drink less than 1 serving of the beverage in the next week. Responses will be averaged to a create a mean intentions score. Response options are on a 1 to 7 scale. Thus, mean scores can range from 1-7, with higher scores indicating higher intentions to limit consumption of these beverages.
Time Frame: Within 30 minutes following completion of ~10-minute shopping task
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sugar-Sweetened Beverage Health Warning Label | Neutral Label
Number analyzed (Participants) | 200 | 200
score on a scale | 5.5 (1.5) | 5.0 (1.7)
Statistical Analysis 1: Comparison: Sugar-Sweetened Beverage Health Warning Label vs Neutral Label; Test type: Superiority; p = 0.005, Regression, Linear — The a priori threshold for statistical significance was < 0.05; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.4, 95% CI 2-sided [0.1 to 0.8]

7. Secondary Outcome: Percent of Participants Who Notice the Trial Labels
Description: Noticing of the trial labels will be measured at post-test using 1 item adapted from Roberto et al. (2016). The item asks participants to indicate whether they noticed the trial labels. Response options are 0 (no) and 1 (yes).
Time Frame: Within 30 minutes following completion of ~10-minute shopping task
Measure: Number; unit: percentage of participants
Arm/Group | Sugar-Sweetened Beverage Health Warning Label | Neutral Label
Number analyzed (Participants) | 200 | 200
percentage of participants | 75.0 | 32.5
Statistical Analysis 1: Comparison: Sugar-Sweetened Beverage Health Warning Label vs Neutral Label; Test type: Superiority; p < 0.001, Regression, Logistic — The a priori threshold for statistical significance was < 0.05; Analyses controlled for overweight/obese status and Hispanic ethnicity, which were unbalanced between treatment arms; Mean Difference (Final Values) = 37, 95% CI 2-sided [32 to 43] — [estimate comment as in outcome 3, analysis 1]

8. Secondary Outcome: Mean Attention Score to the Trial Labels
Description: Attention to the trial labels will be measured at post-test using 2 items adapted from Nonnemaker et al. (2010). The items ask participants to rate their agreement with statements about whether the label grabbed their attention and whether they read and looked closely at the label. Responses will be averaged to create a mean attention score. Responses are on a 1 to 5 scale. Thus, mean scores can range from 1-5, with higher scores indicating higher attention to the labels.
Time Frame: Within 30 minutes following completion of ~10-minute shopping task
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sugar-Sweetened Beverage Health Warning Label | Neutral Label
Number analyzed (Participants) | 200 | 200
score on a scale | 3.1 (1.6) | 1.5 (0.8)
Statistical Analysis 1: Comparison: Sugar-Sweetened Beverage Health Warning Label vs Neutral Label; Test type: Superiority; p < 0.001, Regression, Linear — The a priori threshold for statistical significance was < 0.05; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 1.7, 95% CI 2-sided [1.4 to 1.9]

9. Secondary Outcome: Mean Emotional Reactions Score to Trial Labels
Description: Emotional reactions to the trial labels will be measured at post-test using 6 items adapted from Brewer et al. (2018). The items ask participants to indicate the extent to which trial labels elicited particular emotional reactions (e.g., fear, guilt, disgust). Responses will be averaged to create a mean emotional reactions score. Response options are on a 1 to 5 scale. Thus, mean scores can range from 1-5, with higher scores indicating stronger emotional reactions.
Time Frame: Within 30 minutes following completion of ~10-minute shopping task
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sugar-Sweetened Beverage Health Warning Label | Neutral Label
Number analyzed (Participants) | 200 | 200
score on a scale | 1.5 (0.7) | 1.1 (0.2)
Statistical Analysis 1: Comparison: Sugar-Sweetened Beverage Health Warning Label vs Neutral Label; Test type: Superiority; p < 0.001, Regression, Linear — The a priori threshold for statistical significance was < 0.05; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.4, 95% CI 2-sided [0.3 to 0.5]

10. Secondary Outcome: Mean Cognitive Elaboration Score
Description: Cognitive elaboration will be measured at post-test using 2 items adapted from Moodie, MacKintosh & Hammond (2010) and Fathelrahman et al. (2010). Items ask participants to rate the amount they thought about the information conveyed by the trial label and about the health consequences of consuming beverages with added sugar. Responses will be averaged to create a mean cognitive elaboration score. Response options range from 1 to 5. Thus, mean scores can range from 1-5, with higher scores indicating more elaboration.
Time Frame: Within 30 minutes following completion of ~10-minute shopping task
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sugar-Sweetened Beverage Health Warning Label | Neutral Label
Number analyzed (Participants) | 200 | 200
score on a scale | 2.3 (1.3) | 1.2 (0.6)
Statistical Analysis 1: Comparison: Sugar-Sweetened Beverage Health Warning Label vs Neutral Label; Test type: Superiority; p < 0.001, Regression, Linear — The a priori threshold for statistical significance was < 0.05; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 1.1, 95% CI 2-sided [0.9 to 1.3]

11. Secondary Outcome: Mean Social Interactions About the Labels
Description: Social interactions of the labels will be measured at post-test with a single item adapted from Brewer et al. (2018). Participants will rate the extent to which they are likely to have social interactions about the trial label. Response options are on a 1 to 5 scale. Thus, mean scores can range from 1-5, with higher scores indicating a higher likelihood of having social interactions.
Time Frame: Within 30 minutes following completion of ~10-minute shopping task
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sugar-Sweetened Beverage Health Warning Label | Neutral Label
Number analyzed (Participants) | 200 | 200
score on a scale | 2.2 (1.2) | 1.3 (0.7)
Statistical Analysis 1: Comparison: Sugar-Sweetened Beverage Health Warning Label vs Neutral Label; Test type: Superiority; p < 0.001, Regression, Linear — The a priori threshold for statistical significance was < 0.05; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.9, 95% CI 2-sided [0.7 to 1.1]

12. Secondary Outcome: Mean Perceptions of Added Sugar Score Content in Specific Sugar-sweetened Beverages
Description: Perceptions of added sugar content in specific categories of sugar-sweetened beverages (i.e., soda, fruit drinks, sport drinks/flavored waters, sweetened coffee/tea, and energy drinks) will be measured at post-test using items adapted from Roberto et al. (2016). Items ask participants to rate the amount of added sugar they think is in 1 serving of the beverage. Responses will be averaged to create a mean perceptions of added sugar score. Response options are on a 1 to 4 scale. Thus, mean scores can range from 1-4, with higher scores indicating perceiving higher added sugar content.
Time Frame: Within 30 minutes following completion of ~10-minute shopping task
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sugar-Sweetened Beverage Health Warning Label | Neutral Label
Number analyzed (Participants) | 200 | 200
score on a scale | 3.6 (0.3) | 3.6 (0.3)
Statistical Analysis 1: Comparison: Sugar-Sweetened Beverage Health Warning Label vs Neutral Label; Test type: Superiority; p = 0.055, Regression, Linear — The a priori threshold for statistical significance was < 0.05; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.07, 95% CI 2-sided [-0.001 to 0.13]

13. Secondary Outcome: Mean Attitudes Score Toward Consuming Specific Sugar-sweetened Beverages
Description: Attitudes toward consuming specific sugar-sweetened beverages (i.e., soda, fruit drinks, sport drinks/flavored waters, sweetened coffee/tea, and energy drinks) will be measured at post-test using 5 items adapted from Bollard et al. (2016). Items ask participants to rate how healthy/unhealthy it is for them to consume each beverage category. Responses will be averaged to create an average attitudes score. Response options are on a 1 to 7 scale. Thus, mean scores can range from 1-7, with higher scores indicating more positive attitudes toward consuming these sugar-sweetened beverages.
Time Frame: Within 30 minutes following completion of ~10-minute shopping task
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sugar-Sweetened Beverage Health Warning Label | Neutral Label
Number analyzed (Participants) | 200 | 200
score on a scale | 2.3 (0.8) | 2.4 (0.9)
Statistical Analysis 1: Comparison: Sugar-Sweetened Beverage Health Warning Label vs Neutral Label; Test type: Superiority; p = 0.258, Regression, Linear — The a priori threshold for statistical significance was < 0.05; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.10, 95% CI 2-sided [-0.27 to 0.07]

14. Secondary Outcome: Mean Product Attitudes Score Toward Specific Sugar-sweetened Beverages
Description: Product attitudes toward specific sugar-sweetened beverages (i.e., soda, fruit drinks, sport drinks/flavored waters, sweetened coffee/tea, and energy drinks) will be measured at post-test using 10 items adapted from Bollard et al. (2016). Items ask participants to rate the appeal and the coolness of each beverage category. Responses will be averaged to create a mean product attitude score. Responses are on a 1 to 7 scale. Thus, mean scores can range from 1-7, with higher scores indicating more positive product attitudes toward these sugar-sweetened beverages.
Time Frame: Within 30 minutes following completion of ~10-minute shopping task
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sugar-Sweetened Beverage Health Warning Label | Neutral Label
Number analyzed (Participants) | 200 | 200
score on a scale | 4.1 (1.0) | 4.1 (1.1)
Statistical Analysis 1: Comparison: Sugar-Sweetened Beverage Health Warning Label vs Neutral Label; Test type: Superiority; p = 0.416, Regression, Linear — The a priori threshold for statistical significance was < 0.05; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.09, 95% CI 2-sided [-0.30 to 0.13]

15. Secondary Outcome: Mean Outcome Expectations Score Regarding Consumption of Beverages With Added Sugar
Description: Outcome expectations will be measured at post-test with items adapted from Roberto et al. (2016). Participants will rate the extent to which they expect that consuming beverages with added sugar would increase their risk of negative health outcomes (e.g., tooth decay). Responses will be averaged to a create a mean outcome expectations score. Responses are on a 1 to 7 scale. Thus, mean scores can range from 1-7, with higher scores indicating more negative outcome expectations.
Time Frame: Within 30 minutes following completion of ~10-minute shopping task
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sugar-Sweetened Beverage Health Warning Label | Neutral Label
Number analyzed (Participants) | 200 | 200
score on a scale | 6.2 (0.9) | 6.1 (0.9)
Statistical Analysis 1: Comparison: Sugar-Sweetened Beverage Health Warning Label vs Neutral Label; Test type: Superiority; p = 0.609, Regression, Linear — The a priori threshold for statistical significance was < 0.05; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.05, 95% CI 2-sided [-0.14 to 0.24]

16. Other Pre Specified Outcome: Mean Injunctive Norms Score Regarding Consumption of Beverages With Added Sugar
Description: Injunctive norms will be measured at post-test with items adapted from Zoellner et al. (2012). Items ask participants to rate the extent to which people who are important to them think they should drink less than 1 beverage with added sugar per week, would approve of them drinking less than 1 beverage with added sugar per week, and want them to drink less than 1 beverage with added sugar per week. Responses will be averaged to create a mean injunctive norms score. Responses are on a 1 to 5 scale. Thus, mean scores can range from 1-5, with higher scores indicating higher injunctive norms.
Time Frame: Within 30 minutes following completion of ~10-minute shopping task
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sugar-Sweetened Beverage Health Warning Label | Neutral Label
Number analyzed (Participants) | 200 | 200
score on a scale | 3.8 (0.9) | 3.6 (0.9)
Statistical Analysis 1: Comparison: Sugar-Sweetened Beverage Health Warning Label vs Neutral Label; Test type: Superiority; p = 0.002, Regression, Linear — The a priori threshold for statistical significance was < 0.05; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.3, 95% CI 2-sided [0.1 to 0.5]

17. Other Pre Specified Outcome: Mean Perceived Message Effectiveness of Trial Label
Description: Perceived message effectiveness will be measured at post-test with 1-item adapted from Brewer et al. (2018). Participants will rate the extent to which the trial label would discourage them from drinking beverages with added sugar. Response options are on a 1 to 5 scale. Thus, mean scores can range from 1-5, with higher scores indicating higher perceived effectiveness.
Time Frame: Within 30 minutes following completion of ~10-minute shopping task
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sugar-Sweetened Beverage Health Warning Label | Neutral Label
Number analyzed (Participants) | 200 | 200
score on a scale | 3.3 (1.3) | 1.3 (0.8)
Statistical Analysis 1: Comparison: Sugar-Sweetened Beverage Health Warning Label vs Neutral Label; Test type: Superiority; p < 0.001, Regression, Linear — The a priori threshold for statistical significance was < 0.05; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 2.1, 95% CI 2-sided [1.8 to 2.3]

18. Other Pre Specified Outcome: Mean Support for Sugar-sweetened Beverage Health Warning Labels Score
Description: Support for sugar-sweetened beverage health warning labels will be measured at post-test with 1 item adapted from Brewer et al. (2018). Participants rate their support for a policy that would require health warning labels on sugar-sweetened beverages. Responses are on a 1 to 4 scale. Thus, mean scores can range from 1-4, with higher scores indicating greater support.
Time Frame: Within 30 minutes following completion of ~10-minute shopping task
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sugar-Sweetened Beverage Health Warning Label | Neutral Label
Number analyzed (Participants) | 200 | 200
score on a scale | 3.4 (0.8) | 3.5 (0.7)
Statistical Analysis 1: Comparison: Sugar-Sweetened Beverage Health Warning Label vs Neutral Label; Test type: Superiority; p = 0.311, Regression, Linear — The a priori threshold for statistical significance was < 0.05; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.08, 95% CI 2-sided [-0.23 to 0.07]

19. Other Pre Specified Outcome: Mean Self-efficacy to Limit Consumption of Beverages With Added Sugar Score
Description: Self-efficacy to limit consumption of beverages with added sugar will be measured at post-test with items adapted from Brewer et al. (2018). Items ask participants to rate the extent to which: it would be easy to drink less than 1 beverage with added sugar per week, they have the ability to drink less than 1 beverage with added sugar per week, and they are confident that they could drink less than 1 beverage with added sugar per week. Responses will be averaged to create a mean self-efficacy score. Responses are on a 1 to 5 scale. Thus, mean scores can range from 1-5, with higher scores indicating self-efficacy.
Time Frame: Within 30 minutes following completion of ~10-minute shopping task
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sugar-Sweetened Beverage Health Warning Label | Neutral Label
Number analyzed (Participants) | 200 | 200
score on a scale | 4.2 (1.0) | 4.2 (0.9)
Statistical Analysis 1: Comparison: Sugar-Sweetened Beverage Health Warning Label vs Neutral Label; Test type: Superiority; p = 0.253, Regression, Linear — The a priori threshold for statistical significance was < 0.05; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.11, 95% CI 2-sided [-0.30 to 0.08]

20. Other Pre Specified Outcome: Mean Response Efficacy of Limiting Consumption of Beverages With Added Sugar Score
Description: Response efficacy of limiting consumption of beverages with added sugar will be measured at post-test with items adapted from Brewer et al. (2018). Participants will indicate the extent to which drinking no beverages with added sugar would lower their chances of weight gain, diabetes, tooth decay, and heart disease, and the extent to which drinking no beverages with added sugar would improve their health. Responses are on a 1 to 5 scale. Thus, mean scores can range from 1-5, with higher scores indicating greater response efficacy.
Time Frame: Within 30 minutes following completion of ~10-minute shopping task
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sugar-Sweetened Beverage Health Warning Label | Neutral Label
Number analyzed (Participants) | 200 | 200
score on a scale | 3.9 (0.9) | 4.0 (0.9)
Statistical Analysis 1: Comparison: Sugar-Sweetened Beverage Health Warning Label vs Neutral Label; Test type: Superiority; p = 0.658, Regression, Linear — The a priori threshold for statistical significance was < 0.05; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.04, 95% CI 2-sided [-0.22 to 0.14]

21. Post Hoc Outcome: Mean Number of Calories (kcal) Purchased From Food
Description: Calories from food purchases is defined as the total number of calories from foods in the participant's basket when they complete the shopping task, calculated as the sum of calories/product for all food products. Purchases will be recorded by the experimenter immediately after the participant completes the ~10-minute shopping task.
Time Frame: At completion of ~10-minute shopping task
Measure: Mean (Standard Deviation); unit: kcal
Arm/Group | Sugar-Sweetened Beverage Health Warning Label | Neutral Label
Number analyzed (Participants) | 200 | 200
kcal | 2208.7 (1149.2) | 2259.5 (1069.6)
Statistical Analysis 1: Comparison: Sugar-Sweetened Beverage Health Warning Label vs Neutral Label; Test type: Superiority; p = 0.661, Regression, Linear — The a priori threshold for statistical significance was < 0.05; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -49.5, 95% CI 2-sided [-271.3 to 172.3]

22. Post Hoc Outcome: Mean Number of Calories (kcal) Purchased From Non-sugar-sweetened Beverages
Description: Calories from non-sugar-sweetened beverage purchases is defined as the total number of calories from non-sugar-sweetened beverages in the participant's basket when they complete the shopping task, calculated as the sum of calories/container for all non-sugar-sweetened beverage containers. Purchases will be recorded by the experimenter immediately after the participant completes the ~10-minute shopping task.
Time Frame: At completion of ~10-minute shopping task
Measure: Mean (Standard Deviation); unit: kcal
Arm/Group | Sugar-Sweetened Beverage Health Warning Label | Neutral Label
Number analyzed (Participants) | 200 | 200
kcal | 47.1 (77.2) | 32.9 (63.1)
Statistical Analysis 1: Comparison: Sugar-Sweetened Beverage Health Warning Label vs Neutral Label; Test type: Superiority; p = 0.082, Two-part regression model with robust SE — The a priori threshold for statistical significance was < 0.05; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 12.5, 95% CI 2-sided [-1.6 to 26.6]

ADVERSE EVENTS:
Time Frame: From the time of signing the Informed consent through study task completion, a total of approximately 1 hour.
Arm/Group | Sugar-Sweetened Beverage Health Warning Label | Neutral Label
All-Cause Mortality (participants affected / at risk) | 0/200 | 0/200
Serious Adverse Events (participants affected / at risk) | 0/200 | 0/200
Other Adverse Events (participants affected / at risk) | 0/200 | 0/200

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-30): https://cdn.clinicaltrials.gov/large-docs/37/NCT03511937/Prot_SAP_000.pdf